CLINICAL TRIAL: NCT05440331
Title: Morbidity and Mortality in Operating Room: Surgery and Standardized Communication
Brief Title: Morbidity and Mortality: Surgery and Standardized Transmission in Operating Room
Acronym: HIATUS
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP210992; 2022-A01109-34 (Registry Identifier: IDRCB)
Record Dates: First submitted 2022-06-17; First posted 2022-06-30 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Major Surgery
Keywords: Major surgery; Morbility; Mortality; Training in peroperative; Handover; Anaesthetist; Nurse anaesthetist

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Experimental group: Experimental group with training after randomization immediately
  Interventions: Other: Training with AnesList©
- Control group with delayed training: Control group with training: the training will delayed from time of randomization
  Interventions: Other: Training with AnesList©
- Control group without training: Control group without training

INTERVENTIONS:
Other: Training with AnesList© — Training with AnesList© as tool
  Groups: Control group with delayed training; Experimental group

SUMMARY:
The primary objective of the study is to evaluate the efficacy of standard handover with AnesList© between physician anesthesists in operating room, for a complete transmission for a patient, on the occurence of event as death, serious complications or rehospitalization in month of postoperative after major surgery.

DETAILED DESCRIPTION:
The secondary objectives are:

* to analysis the impact of the transmission on:

  1. the occurence of different events: re-hospitalization, serious complications, death at one month;
  2. the duration of initial ICU stay and of hospitalization;
  3. the duration of the transmission;
  4. the quality of the transmission by the physician leaving operating room.
* to evaluate the condition of the transmission
* to study the persistence of the use of the AnesList© at 6 months after the end of inclusions in the center
* to evaluate the satisfaction on AnesList© and on the training with the tool and the obstacles of its utilization
* to evaluate the morbility-mortality in the centers of the centers before, during and 6 months after the beginning of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged > 18 years;
* Patients with score ASA I-IV;
* Requiring urgent or planned surgery;
* Major surgery (duration of surgery > 2 hours, requiring a hospital stay of at least 1 night): orthopedics, cardiac, vascular, thoracic, visceral, ENT, plastic surgery;
* Handover between two anesthesists defined as a definitive relay between one physician anaesthesist and another in operating room;
* Intensive care anesthesists and nurse anaesthetist working in investigator center during the study;
* Affiliated to a social security system;
* No-opposition to participating to the study.

Exclusion Criteria:

* Transmission between physician anaesthesist and nurse anaesthetist;
* Medical transmission occurs out of anesthesia care out of operating room;
* Medical transmission occurs in transitory manner (for example: coffee time, lunch time);
* Patients enrolled in an another ongoing study of surgical intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients requiring urgent or planned major surgery (duration of surgery > 2 hours, requiring a hospital stay of at least 1 night): orthopedics, cardiac, vascular, thoracic, visceral, ENT, plastic surgery; with handover between two anesthesists defined as a definitive relay between one physician anaesthesist and another in operating room; Intensive care anesthesists and nurse anaesthetist working in investigator center during the study.
Sampling Method: Probability Sample
Enrollment: 1120 (Estimated)
Dates: Start 2023-09-08 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
The occurence of adverse events | at 1 month
  Death, serious complications and re-hospitalization will be noted in order to evaluate the efficacy of standardized transmission with AnesList©.

SECONDARY OUTCOMES:
The duration of ICU stay | through study completion, an average of 18 months
  The length of initial ICU stay will be noted.
The duration of hospitalization | through study completion, an average of 18 months
  The length of initial hospitalization will be noted.
Evaluate of the condition of transmission | through study completion, an average of 18 months
  By the presence or intervention of anaesthetics-nurse, recorded or not the transmission in medical files.
Utilization of the AnesList© by anaesthesists at 6 months | at 6 months
  Only for intervention group: use on cell phone or with printed form: the use will be noted.
Quality of medical transmission | through study completion, an average of 18 months
  Scale will be noted by anaesthesists between 0 and 22: 20% of recorded transmission will be noted.
Interaction with study nurse | through study completion, an average of 18 months
  The study nurse will evaluate the existence and composite of the interaction between the anesthesist who receiving the transmission and the nurse.
Morbi-mortality | through study completion, an average of 18 months
  The method of chronological series will be used to analysis the morbi-mortality in investigator center.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique FLETCHER, MD, PhD, Principal Investigator — Department of Anesthesia and Intensive Care - Ambroise Paré Hospital - APHP; Aicha KASSOUL, MD, Study Director — Department of Anesthesia and Intensive Care - Ambroise Paré Hospital - APHP
Locations (1):
- Department of Anesthesia and Intensive Care - Ambroise Paré Hospital - APHP, Boulogne-Billancourt, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sedgwick P, Greenwood N. Understanding the Hawthorne effect. BMJ. 2015 Sep 4;351:h4672. doi: 10.1136/bmj.h4672. No abstract available. PMID 26341898
- [Background] Jullia M, Tronet A, Fraumar F, Minville V, Fourcade O, Alacoque X, LeManach Y, Kurrek MM. Training in intraoperative handover and display of a checklist improve communication during transfer of care: An interventional cohort study of anaesthesia residents and nurse anaesthetists. Eur J Anaesthesiol. 2017 Jul;34(7):471-476. doi: 10.1097/EJA.0000000000000636. PMID 28437261
- [Background] Haynes AB, Weiser TG, Berry WR, Lipsitz SR, Breizat AH, Dellinger EP, Herbosa T, Joseph S, Kibatala PL, Lapitan MC, Merry AF, Moorthy K, Reznick RK, Taylor B, Gawande AA; Safe Surgery Saves Lives Study Group. A surgical safety checklist to reduce morbidity and mortality in a global population. N Engl J Med. 2009 Jan 29;360(5):491-9. doi: 10.1056/NEJMsa0810119. Epub 2009 Jan 14. PMID 19144931